CLINICAL TRIAL: NCT02237547
Title: Safety and Feasibility Study of Cell Therapy in Treatment of Spinal Cord Injury
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrollment.
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNEI-2014-TBS-UCMSC-SCI001
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; mesenchymal; bone marrow; mononuclear cells; stem cells; umbilical cord
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV and IT UC-MSC and BMMC (Experimental): Intravenous and intrathecal human umbilical cord tissue-derived mesenchymal stem cells and bone marrow mononuclear cells
  Interventions: Biological: Intravenous and intrathecal human umbilical cord tissue-derived mesenchymal stem cells and bone marrow mononuclear cells

INTERVENTIONS:
Biological: Intravenous and intrathecal human umbilical cord tissue-derived mesenchymal stem cells and bone marrow mononuclear cells

SUMMARY:
Human Umbilical Cord-derived Mesenchymal Stem Cells (UC-MSC) and Bone Marrow Mononuclear Cells (BMMC) from the patient injected into the spinal fluid intrathecally and injected intravenously (IV) is a safe and therapeutic procedure for spinal cord injury (SCI) patients.

DETAILED DESCRIPTION:
The proposed study will assess primary safety and secondary efficacy endpoints of autologous bone marrow mononuclear cells and allogeneic human umbilical cord-derived mesenchymal stem cells administered to 20 male and female subjects between ages of 18-50 with spinal cord injury. These cells will be administered intrathecally and intravenously multiple times over the course of one month.

The primary objective is freedom from treatment-associated adverse events at 3 and 12 months post-treatment. Secondary objective will be efficacy at baseline, 3 months and 12 months and will be quantified based on the following: American Spinal Cord Injury Association (ASIA) classification and the Frankel Scale.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between age 18 and 50
* Paraplegics and quadriplegics with complete or incomplete spinal cord injuries.
* Willingness to undergo bone marrow derived autologous cell therapy.
* Ability and willingness to make regular visits to hospital and follow ups during the protocol procedure and comply with all medical instructions
* Traumatic Injury of spinal cord with complete or partial damage by Magnetic Resonance Imaging (MRI) and injury level below C4
* ASIA impairment scale from A - C
* Must have proof of health insurance in country of residence.
* Signed informed consent

Exclusion Criteria:

* Pre- existing or current systemic disease such as lung, liver (exception: history of uncomplicated hepatitis A), gastrointestinal, cardiac, Human Immunodeficiency Virus (HIV)
* History of life threatening allergic- or immune-mediated reaction
* Hemodynamic instability
* Peripheral muscular dystrophy
* Lactating or pregnant woman
* Women capable of childbearing unwilling to use multiple forms of contraception
* Alcohol drug abuse /dependence
* Positive test result for hepatitis A and Hepatitis B OR C
* Major-traumatic brain injury and psychiatric illness
* Open injuries
* Active infectious diseases
* Life expectancy of less than one year due to terminal condition
* Neurodegenerative diseases
* Primary hematologic diseases
* Any of the following medications that cannot be discontinued one week prior to the first stem cell administration and throughout the course of treatment. (1 week before visit 2 through one week after visit 12)

  * Antibiotics
  * Antifungals
  * Antivirals
  * Blood thinners (to avoid bleeding risk during bone marrow aspiration and IT procedures)
  * High doses of Vitamin D or fish oils (since these might prolong bleeding times)
* Bone reflecting increased risk for spinal puncture
* Hepatic dysfunction
* Other medical complications that contraindicate surgery, including major respiratory complications
* Participation in another clinical trial
* Coagulopathies
* Uncorrected coagulopathy during the baseline period defined as: International Normalized Ratio (INR) > 1.4; Partial Thromboplastin Time (PTT) > 35 sec; Platelet Count (PLT) < 100,000.
* Pre-injury history of seizure disorder and/or neurological impairment where participation in age-appropriate pain rating scales would not be practical or possible
* Subject does not sign informed consent form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 12 weeks, 52 weeks
  12 and 52 weeks after final treatment

SECONDARY OUTCOMES:
Number of subjects with a change in American Spinal Injury Association (ASIA) score from baseline | 12 weeks, 52 weeks
  12 and 52 weeks after final treatment
Number of subjects with a change in Frankel Scale score from baseline | 12 weeks, 52 weeks
  12 and 52 weeks from final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Novarro, MD, Principal Investigator
Locations (1):
- Stem Cell Institute, Panama City, Panama